CLINICAL TRIAL: NCT03001349
Title: An Expanded Access Imaging of Neuroendocrine Tumors Using 68Ga-DOTA-TOC
Brief Title: 68Ga-DOTA-TOC PET/CT in Imaging Participants With Neuroendocrine Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0030; NCI-2018-01894 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0030 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Meningioma; Metastatic Well Differentiated Neuroendocrine Neoplasm; Multiple Endocrine Neoplasia Type 1; Neuroendocrine Neoplasm; Somatostatin Positive Neoplastic Cells Present; Von Hippel-Lindau Syndrome
MeSH Terms: conditions — Meningioma; Multiple Endocrine Neoplasia Type 1; Neuroendocrine Tumors; von Hippel-Lindau Disease | interventions — gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (gallium Ga 68-edotreotide, PET/CT) (Experimental): Participants receive gallium Ga 68-edotreotide intravenously. After 1 hour, participants undergo PET/CT scan over 60 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-Edotreotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Gallium Ga 68-Edotreotide — Given IV
  Other Names: 68Ga-DOTA-d-Phe1-Tyr3-octreotide; 68Ga-DOTA-TOC; EDOTREOTIDE GALLIUM GA-68; Ga-68 DOTA0-Tyr3-octreotide; Ga-68 DOTATOC; Ga-68-DOTA-TOC; Ga-68-DOTA-Tyr(3)-octreotide; Gallium Ga 68-DOTATOC
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well gallium Ga 68-edotreotide (68Ga-DOTA-TOC) positron emission tomography (PET)/computer tomography (CT) works in imaging participants with neuroendocrine tumors. 68Ga-DOTA-TOC is used as a tracer chemical during PET/CT scans. Diagnostic procedures, such as 68Ga-DOTA-TOC PET/CT, may help find and diagnose neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To substitute 68Ga-DOTATOC for 111In-pentetreotide on an expanded access basis, in tumor imaging for study subjects, where the care provider believes that somatostatin imaging is clinically indicated, until such time as 68Ga-DOTATOC becomes commercially available.

SECONDARY OBJECTIVES:

I. To gain experience in the utility of 68Ga-DOTATOC in the management of neuroendocrine tumors at The University of Texas M.D. Anderson Cancer Center (MDACC).

II. To acquire proficiency in generating 68Ga-DOTATOC for human use at MDACC.

OUTLINE:

Participants receive gallium Ga 68-edotreotide intravenously. After 1 hour, participants undergo PET/CT scan over 60 minutes.

After completion of study, participants are followed up at 24 hours or within 72 hours, and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the subject, or the legally authorized representative (LAR), if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable, to understand, and the willingness to sign, a written informed consent
* All participants must meet one of the following:

  * Patients diagnosed or suspected to have neuroendocrine tumors (NET), who require 111In-pentetreotide imaging for clinical indications
  * Subjects with a high risk of NET because of familial predisposition, and also have clinical findings which require radiolabeled somatostatin imaging
  * Other somatostatin-positive tumors for which 111In-pentetreotide has been used successfully, such as adult meningiomas
  * Patients with suspected neuroendocrine tumor, unknown primary NET, metastatic NET, or other tumors, such as meningiomas, in whom the primary physician considers somatostatin imaging to be clinically indicated
  * Other NET subjects, whether asymptomatic or symptomatic, sporadic or familial, such as Von Hippel-Lindau syndrome (VHL) and multiple endocrine neoplasia type 1 (MEN1), will also be included

Exclusion Criteria:

* Pregnant women are excluded from this study because the effects of 68Ga-DOTATOC in pregnancy are not known; exceptions may be granted only if the expected risk outweighs the benefit, in the clinical opinion of the attending physician. Pregnancy testing will follow MD Anderson procedure for diagnostic reagents. Self-reporting is used to assess pregnancy status. If the subject is unsure about her status, a urine or serum pregnancy test will be performed before inclusion
* Lactating women are excluded if patient is unwilling to suspend lactation for at least one day following the administration of 68Ga-DOTATOC to the mother, because of the unknown but potential risk for adverse events in nursing infants secondary to administration of the radionuclide to a lactating woman
* Subjects with known contraindications to the use of 111In-pentetreotide
* Known severe allergy or hypersensitivity to oral contrast precludes administration of oral contrast only
* Patients with a body weight of 400 pounds or more, or a body mass index (BMI) which precludes their entry into the bore of the PET/CT scanner, because of the resulting probable compromise in image quality with CT, PET/CT and magnetic resonance imaging (MRI)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator may significantly interfere with study compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  As measured by National Cancer Institute Common Terminology Criteria for Adverse Events version 4. Traceable toxicity/safety data will be assessed. Adverse events and vital signs will be monitored and described with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Homer A Macapinlac, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org